CLINICAL TRIAL: NCT03711539
Title: Lifetime Endurance Exercise to Prevent Coronary Artery Disease. A Comparison With Late-onset Endurance Training and a Sedentary Lifestyle
Brief Title: Lifetime Endurance Exercise to Prevent Coronary Artery Disease
Acronym: MASTER@HEART
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University Hospital, Antwerp (Other); Jessa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: S61336
Record Dates: First submitted 2018-10-17; First posted 2018-10-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease; Physical Activity; Lifestyle
Keywords: Endurance Exercise; Coronary Artery Disease; Atrial Fibrillation; Myocardial Fibrosis; Coronary CT
MeSH Terms: conditions — Coronary Artery Disease; Motor Activity; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lifelong Endurance Athletes: i) Athletes who have initiated endurance sports activities at regional, national or international level before the age of 30 years. Sports include triathlon, cycling, distance running (1500 metres and longer) and rowing. ii) Aged 45-70 years. iii) Involved in competition and high-level training: more than 10 hours per week for cyclists and triathletes or more than 6 hours per week for runners and rowers. Subjects will be excluded if: i) they have a history of smoking (> 5 pack years) or diabetes, ii) had been diagnosed with a cardiopulmonary disorder prior to inclusion.
- Late-onset Endurance Athletes: i) Athletes who have initiated endurance sports activities at regional, national or international level after the age of 30 years. Sports include triathlon, cycling, distance running (1500 metres and longer) and rowing. ii) Aged 45-70 years. iii) Involved in competition and high-level training: more than 10 hours per week for cyclists and triathletes or more than 6 hours per week for runners and rowers. Subjects will be excluded if: i) they have a history of smoking (> 5 pack years) or diabetes, ii) they have a history of smoking (> 5 pack years) or diabetes, ii) had been diagnosed with a cardiopulmonary disorder prior to inclusion.
- Healthy Non-athletes: Healthy non-athletes will be recruited from subjects seen in the outpatient clinic for a work-related medical check-up, from university alumni and from multisports organisations. Subjects will be excluded if they: i) had been involved in regular sports practice more than >3 hours / week, ii) have a history of smoking (> 5 pack years) or diabetes, or iii) had been diagnosed with a cardiopulmonary disorder prior to inclusion. Participation in regular sports with a low dynamic component (e.g. billiards, darts or bowling) >3 hours /week is allowed.

SUMMARY:
The primary objective of the Master@Heart Trial is to investigate whether lifelong endurance exercise reduces the incidence of non-calcified plaques (both mixed and soft plaques) as compared to late-onset endurance exercise and a non-athletic lifestyle.

DETAILED DESCRIPTION:
Cardiovascular disease remains the leading cause of death in Europe and is strongly related to a sedentary lifestyle combined with inadequate dietary habits and the prevalence of smoking. In parallel with this modern inactivity pandemic, the past 2 decades we have also witnessed an increase in the number of middle-aged and older individuals engaging in competitive sports and mass exercise events, such as marathon-running and cycling events. This increasing popularity of endurance sports implies that a greater proportion of individuals participating in high-intensity sport will have a higher cardiovascular risk profile. Coronary artery disease is by far the most common cause of sudden cardiac death in senior athletes, accounting for >75% of all cardiac deaths during exercise. Each case of sudden cardiac death is always a dramatic event and is often widely publicized in the media, thereby raising issues and questions regarding the safety of intense sports participation. Debate and uncertainty persist with much speculation filling the space left by an incomplete understanding of the exercise dose-response relationship. In view of the importance of exercise for healthy ageing, it is important to identify and eliminate any adverse associations with exercise so that everyone can enjoy the benefits of exercise. Until present, no studies have compared the 'standard of care,' which includes a healthy diet, abstinence from smoking, and regular moderate exercise, with and without the addition of larger doses of endurance exercise. Furthermore, it remains unknown whether the age of onset of endurance training influences its potential preventive and adverse effects.

Until present, no studies have compared the 'standard of care,' which includes a healthy diet, abstinence from smoking, and regular moderate exercise, with and without the addition of long-term endurance exercise. In this multicentre project we will investigate the beneficial effects of long-term endurance exercise for the prevention of coronary and carotid artery disease and its potential adverse effects, such as an increased incidence of atrial fibrillation and myocardial fibrosis. We will recruit 3 age-matched cross-sectional cohorts: (1) lifelong endurance athletes engaged in regular endurance sports practice since the age of 30 years, (2) late-onset endurance athletes who have initiated endurance sports activities after the age of 30 years and (3) non-athletic individuals. Only male subjects will be included given the much lower prevalence of ischemic heart disease amongst female athletes.

ELIGIBILITY:
Inclusion Criteria:

* Lifelong endurance athletes:

  * Initiation of endurance sports before the age of 30 years
  * Activities at regional, national or international level
  * Sports: triathlon, cycling, distance running (1500 metres and longer) and rowing
  * Aged 45-70 years
  * Involved in competition and high-level training:

    * more than 10 hours per week for cyclists and triathletes
    * more than 6 hours per week for runners and rowers.
* Late-onset endurance athletes:

  * Initiation of endurance sports after the age of 30 years and at least 6 months ago
  * Activities at regional, national or international level
  * Sports: triathlon, cycling, distance running (1500 metres and longer) and rowing
  * Aged 45-70 years
  * Involved in competition and high-level training:

    * more than 10 hours per week for cyclists and triathletes
    * more than 6 hours per week for runners and rowers.
* Healthy non-athletes

  * subjects seen in the outpatient clinic for a work-related medical check-up
  * university alumni
  * subjects from multisports organisations
  * history of regular sports practice <3 hours /week
  * participation in regular sports with a low dynamic component (e.g. billiards, darts or bowling) >3 hours /week is allowed

Exclusion Criteria:

* history of smoking (> 5 pack years)
* history of diabetes
* diagnosis of cardiopulmonary disorder prior to inclusion
* medical treatment for arterial hypertension or hypercholesterolemia

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1: Lifelong endurance athletes. Inclusions: Athletes who have initiated endurance sports activities at regional, national or international level before the age of 30 years. Sports include triathlon, cycling, distance running (1500 metres and longer) and rowing.
  Cohort 2: Late-onset endurance athletes. Athletes who have initiated endurance sports activities at regional, national or international level after the age of 30 years. Sports include triathlon, cycling, distance running (1500 metres and longer) and rowing.
  Cohort 3: Healthy non-athletes will be recruited from subjects seen in the outpatient clinic for a work-related medical check-up, from university alumni and from multisports organisations. Participation in regular sports with a low dynamic component (e.g. billiards, darts or bowling) >3 hours /week is allowed.
Sampling Method: Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2018-10-18 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Non-calcified Plaques | 2 years
  Incidence of non-calcified plaques (both mixed and soft plaques) assessed by Coronary CT in lifelong endurance athletes as compared to late-onset endurance athletes and non-athletic subjects.

SECONDARY OUTCOMES:
Incidence of Atrial Fibrillation | 4 years
  To assess the association between the (a) amount and (b) starting age of lifelong endurance sports and atrial fibrillation assessed by Holter monitoring
Prevalence of Myocardial Fibrosis | 2 years
  To assess the association between the (a) amount and (b) starting age of lifelong endurance sports and myocardial fibrosis assessed by cardiac magnetic resonance imaging

OTHER OUTCOMES:
Arterial Stiffness | 2 years
  To assess arterial stiffness by Applanation Tonometry in lifelong endurance athletes versus late-onset athletes and non-athletic individuals.
Carotid Intima Thickness | 2 years
  To assess carotid intima thickness by Doppler Ultrasound in lifelong endurance athletes versus late-onset athletes and non-athletic individuals.
Left Ventricular Diastolic Function | 2 years
  To assess left ventricular diastolic function by echocardiography in lifelong endurance athletes versus late-onset athletes and non-athletic individuals.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - University Hospital, Antwerpen, Edegem
  - Jessa Hospital, Hasselt
  - UZLeuven, Leuven

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Janssens K, Foulkes SJ, Mitchell AM, Dausin C, Van Soest S, Spencer L, Rowe SJ, D'Ambrosio P, Elliott AD, Van Puyvelde T, Parr EB, Willems R, Heidbuchel H, Claessen G, La Gerche A. Blood pressure response to graded bicycle exercise in males and females across the age and fitness spectrum. Eur J Prev Cardiol. 2025 Jan 6;32(1):43-51. doi: 10.1093/eurjpc/zwae262. PMID 39116385
- [Derived] De Bosscher R, Dausin C, Claus P, Bogaert J, Dymarkowski S, Goetschalckx K, Ghekiere O, Belmans A, Van De Heyning CM, Van Herck P, Paelinck B, El Addouli H, La Gerche A, Herbots L, Heidbuchel H, Willems R, Claessen G. Endurance exercise and the risk of cardiovascular pathology in men: a comparison between lifelong and late-onset endurance training and a non-athletic lifestyle - rationale and design of the Master@Heart study, a prospective cohort trial. BMJ Open Sport Exerc Med. 2021 Apr 16;7(2):e001048. doi: 10.1136/bmjsem-2021-001048. eCollection 2021. PMID 33927885